CLINICAL TRIAL: NCT01052402
Title: A Phase 1/2 Study to Assess the Safety and Immunogenicity of a Vero Cell-Derived Whole Virus H5N1 Influenza Vaccine in Healthy Infants, Children and Adolescents Aged 6 Months to 17 Years
Brief Title: Safety and Immunogenicity Study of a H5N1 Influenza Vaccine (Vero Cell-Derived, Whole Virus) in Healthy Infants, Children and Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 810706
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2012-11

CONDITIONS: Influenza, Avian
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose A (Experimental): Two intramuscular injections (21 days apart, i.e. Days 0 and 21) of H5N1 Influenza Vaccine (Dose A) followed by a heterologous booster vaccination (Dose A) on Day 360
  Interventions: Biological: H5N1 Influenza Vaccine (Whole Virion, Vero Cell-Derived, Inactivated), non-adjuvanted formulation
- Dose B (Experimental): Two intramuscular injections (21 days apart, i.e. Days 0 and 21) of H5N1 Influenza Vaccine (Dose B) followed by a heterologous booster vaccination (Dose B) on Day 360
  Interventions: Biological: H5N1 Influenza Vaccine (Whole Virion, Vero Cell-Derived, Inactivated), non-adjuvanted formulation

INTERVENTIONS:
Biological: H5N1 Influenza Vaccine (Whole Virion, Vero Cell-Derived, Inactivated), non-adjuvanted formulation — Two vaccinations, 21 days apart, followed by a heterologous booster vaccination on Day 360

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity (i.e. primary immune response, immunogenicity of two different doses, antibody persistence 360 days after the first vaccination, immune response to a heterologous booster given on Day 360) of a Vero cell-derived whole virus H5N1 influenza vaccine in healthy infants, children and adolescents aged 6 months to 17 years.

ELIGIBILITY:
Inclusion Criteria:

* 9 to 17 years of age on the day of screening (for Stratum A only)
* 3 to 8 years of age on the day of screening (for Stratum B only)
* 6 to 35 months of age on the day of screening (for Stratum C only)
* Subject who were born at full term of pregnancy (>= 37 weeks) with a birth weight >= 2 kg (for Stratum C only)
* Subjects and/or their parents/legal guardians understand the nature and procedures of the study and agree to its provisions
* Subjects´ parents/legal guardians provide written consent for participation according to national law. In case the parents/legal guardians are illiterate, the informed consent is also to be signed by an independent witness
* Written assent according to subjects´ age and capacity of understanding
* Subjects who are generally healthy, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination
* Subjects who are physically and mentally capable of participating in the study and follow its procedures
* Subjects and/or their parents/legal guardians agree to keep a daily record of symptoms for the duration of the study
* If subjects are female of childbearing potential - have a negative urine pregnancy test result within 24 hours prior to the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* History of exposure to H5N1 virus or a history of vaccination with an H5N1 influenza vaccine
* High risk of contracting H5N1 influenza infection (e.g. contact with poultry);
* Subjects who currently have or have a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Inherited or acquired immunodeficiency
* Subjects who have a disease or are currently undergoing a form of treatment or were undergoing a form of treatment within 30 days prior to study entry that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs.
* History of severe allergic reactions or anaphylaxis
* Rash, dermatological condition or tattoos which may interfere with injection site reaction rating
* Subjects who have received a blood transfusion or immunoglobulins within 90 days prior to study entry
* Subjects who have received any live vaccine within 4 weeks or inactivated vaccine within 2 weeks prior to vaccination in this study
* Functional or surgical asplenia
* Subjects with a known or suspected problem with alcohol or drug abuse
* Subjects who were administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* Dependent relationship with the study site personnel. Dependent relationships include close relatives (i.e., children, siblings).
* If female: subjects wo are pregnant or lactating

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 684 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of systemic reactions until 7 days after the first vaccination | 7 days
Rate of subjects with antibody response to the vaccine strain associated with protection 21 days after the second vaccination defined as titer measured by Microneutralization test >= 1:20. | 42 days

SECONDARY OUTCOMES:
Frequency and severity of systemic and injection site reactions until 21 days after the first, second and booster vaccination | Day 21, 42 and 381
Fever, malaise or shivering (in children and adolescents aged 3 to 17 years) and fever and irritability (in infants and young children aged 6 to 35 months) with onset within 7 days after the first, second and booster vaccination | Day 21, 42 and 381
Adverse events observed during the entire study period | Throughout entire study period
Antibody response associated with protection 21 days after the first and second vaccination, and again at 360 days after the first vaccination and 21 days after the booster vaccination | Day 21, 42, 360 and 381
  Antibody response defined as Hemagglutination Inhibition Antibody (HIA) titer >= 1:40 or Single Radial Hemolysis (SRH) area >= 25 mm2, and as measured by Microneutralization (MN) test >= 1:20
Fold increase of antibody response 21 days after first and second vaccination as compared to baseline, and again at 21 days after the booster vaccination as compared to before the booster vaccination | Day 21, 42, 360 and 381
  Measured by MN, HI and SRH assay
Seroconversion 21 days after the first and second vaccination and at 21 days after the booster vaccination | Day 21, 42 and 381
  Measured by MN, HI and SRH assay

CONTACTS AND LOCATIONS:
Overall Officials: BioScience Investigator, MD, Study Director — Baxter Innovations GmbH
Locations (20):
- Princess Margaret Hospital for Children, Subiaco, Australia
- Finland (10):
  - Tampere University, Espoo Vaccine Research (Tampereen Yliopisto, Espoon Rokotetutkimus), Espoo
  - South Helsinki Vaccine Research Clinic (Etelä-Helsingin Rokotetutkimusklinikka), Helsinki
  - Kokkola Vaccine Research Clinic (Kokkolan Rokotetutkimusklinikka), Kokkola
  - Kuopion Vaccine Research Clinic, Kuopio
  - Oulu Vacine Research Clinic (Oulun Rokotetutkimusklinikka), Oulu
  - Porin Vaccine Research Clinic, Pori
  - University of Tampere, Seinäjoki Vaccine Research Clinic (Tampereen Yliopisto, Seinajoen Rokotetutkimusklinikka), Seinäjoki
  - Tampere Vacine Research Clinic (Tampereen Rokotetutkimusklinikka), Tampere
  - Turku Vaccine Research Clinic (Turun Rokotetutkimusklinikka), Turku
  - University of Tampere, Vantaa East Vaccine Research Clinic (Itä Vantaan Rokotetutkimusklinikka), Vantaa
- Singapore (2):
  - The Children´s Medical Institute, Singapore
  - Mount Elizabeth Medical Centre, The Child and Allergy Clinic, Singapore
- Spain (7):
  - Centro de Salud de Paiporta, Paiporta
  - Instituto Hispalense de Pediatria, Pediatría - IHP1, Seville
  - Centro de Salud Malvarrosa, Valencia
  - Centro de Salud Serreria II, Valencia
  - Centro de Salud Trafalgar, Valencia
  - Centro de Salud de Catarroja, Valencia
  - Centro de Salud Quart de Poblet, Valencia

REFERENCES:
- [Derived] van der Velden MV, Fritz R, Pollabauer EM, Portsmouth D, Howard MK, Kreil TR, Dvorak T, Fritsch S, Vesikari T, Diez-Domingo J, Richmond P, Lee BW, Kistner O, Ehrlich HJ, Barrett PN, Aichinger G. Safety and immunogenicity of a vero cell culture-derived whole-virus influenza A(H5N1) vaccine in a pediatric population. J Infect Dis. 2014 Jan 1;209(1):12-23. doi: 10.1093/infdis/jit498. Epub 2013 Sep 16. PMID 24041789